CLINICAL TRIAL: NCT03474159
Title: Evaluation of Aortic Stiffness as a Prognostic Indicator of Aortic Dilatation in Patients With Bicuspid Aortic Valve (BAV) by Multimodal Imaging (MRI, Echocardiography and Ultrafast Ultrasound Imaging)
Brief Title: Evaluation of Aortic Stiffness as a Prognostic Indicator of Aortic Dilatation in Patients With Bicuspid Aortic Valve by Multimodal Imaging
Acronym: IRM-BAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-08
Record Dates: First submitted 2018-02-23; First posted 2018-03-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Bicuspid Aortic Valve
Keywords: Bicuspid aortic valve; aortic aneurysm; stiffness; Pulse wave velocity
MeSH Terms: conditions — Bicuspid Aortic Valve Disease; Aortic Aneurysm | interventions — Magnetic Resonance Imaging; Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Other): patients with Bicuspid aortic valve (defined using the Sievers classification) and confirmed with either Transthoracic Echocardiography, computed tomography, or Magnetic Resonance Imaging Carotid pulse rate measured on carotid arteries by UF
  Interventions: Device: Magnetic Resonance Imaging; Device: Transthoracic echocardiography; Device: Echography UltraFast

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Aortic distensibility measured in MRI at the Valsalva sinus and at the ascending tubular aortic level
  Other Names: MRI
Device: Transthoracic echocardiography — Aortic distensibility measured in TTE of the same segments in TM and in B mode
  Other Names: TTE
Device: Echography UltraFast — Carotid pulse rate measured on carotid arteries by UF
  Other Names: UF

SUMMARY:
The objective is the development and validation of morphological markers informative of aortic dilatation in order to improve the precision of the risk of aneurysm of the thoracic aorta and of acute aortic syndrome for patients with bicuspid aortic valve (BAV).

The primary objective of this study is to demonstrate a correlation between the aortic local pulse wave velocity (PWV) measured with MRI and the progression of the thoracic aorta diameters measured by MRI after a follow-up of 2 years.

DETAILED DESCRIPTION:
Background Bicuspid Aortic Valve (BAV) is the most common congenital heart defect with prevalence around 1 to 2% of the general population . It is defined by the presence of two functional cusps with less than three parallel zones of apposition between the cusps. This different valve's morphology is associated with a spectrum of valvular (aortic stenosis and insufficiency) and aortic complications (aneurysm and dissection). Indeed, the valvular abnormality is associated with changes in the aortic arch with an increase in the incidence of ascending aortic aneurysm unrelated to valvular functional impairment. The mechanisms responsible for aortic involvement are still incompletely understood but combine, in varying proportions, a constitutional fragility (linked to a common embryological origin of the aortic valve and the aortic arch) and to the haemodynamic modifications, generated by the specific morphology of BAV .

Current risk prediction of aneurysm development is currently performed only with the ascending aortic diameter, associated with history of aortic coarctation and familial history of dissection. Moreover, aortic dilatation may occur after aortic valve replacement alone, necessitating a second intervention, with a higher surgical risk. Improvement of the aortopathy evaluation is therefore a major stake in the evaluation of the BAV patient.

Studies of the biomechanical properties of the BAV aortic wall converge towards an increase in arterial stiffness as well as in other elastopathies such as Marfan's disease. Thus, measurements of aortic distensibility in trans-thoracic echocardiography (TTE) or MRI, or the measurement of the Pulse Wave Velocity (PWV) are significantly different case of BAV compared to the general population. However, no prospective study has demonstrated the prognostic role of these morphological biomarkers in the prediction of aortic dilation.

From a biomechanical point of view, the vessel's rupture appears when the mechanical stress applied to the wall exceeds the material resistance properties. The aortic resistance evaluation requires the use of different imaging modalities which propose the measurement of stiffness parameters. Circumferential stiffness (with TTE or MRI) can be evaluated by measuring the distensibility. In addition, longitudinal stiffness can be evaluated by measuring the local PWV.

We aim at better defining the vascular involvement of BAV patients by determining the prognostic role of functional parameters as non-invasive predictive factors for aortic dilation.

Hypothesis:

1.Main hypothesis The main hypothesis is that the progression of aortic dilation is dependent on the longitudinal and circumferential aortic stiffness in case of BAV.

The investigators will therefore try to demonstrate a correlation between the local PWV measurements in MRI, combined with a simultaneous measurement of the non-invasive central pressure (SphygmoCor XCEL®, Atcor Medical ©), with the segmental aortic size progression. The investigators hope to define new biomarkers aortic dilation prediction.

1.Secondary hypothesis

* The measurement of the local PWV of the common carotid artery, measured with UF, is correlated with the progression of the aortic dilation.
* The measurement of aortic distensibility at the Valsalva sinus and ascending tubular aortic levels, measured in TTE or MRI, correlates with the progression of aortic dilation.

Originality and innovative aspects - Prospective evaluation of the different aortic segments dilatation in case of BAV: Few studies have prospectively evaluated the aortic dilation progression in BAV. There are currently no prognostic markers of dilatation validated in this group.

- Use of aortic MRI combined with central pressure measurement as a prognostic evaluation tool for aortopathy associated with BAV: Following the development of 4D MRI in cardiovascular imaging, evaluation of the aorta is possible by studying both the wall's movements during the cardiac cycle and the wall shear stress evaluation. This makes possible to obtain, at each part of the thoracic aorta, measures of circumferential distensibility, local PWV, and shear stress.

Coupling these two imaging modalities is particularly interesting in the aortic evaluation of BAV due to the involvement of the flow changes in aortic stiffness.

- Use of the common carotid artery stiffness as a prognostic evaluation tool for aortopathy associated with BAV independently of the aortic diameter Due to the common embryological origin of aorta and the common carotid arteries, aortopathy associated with BAV is associated with an increase in of the common carotid arteries stiffness.

The evaluation of the carotid artery will therefore help to evaluate the correlation between carotid rigidity and progression of aortic dilation.

- Evaluation of the local PWV as carotid stiffness biomarker Ultrasound analysis will also be innovative, with the use of a fine ultrasonic method with very high frame rate (more than 10,000 images per second) developed by the Langevin Institute (Mathias Fink, Michael Tanter and Mathieu Pernot). The collaboration between the Langevin Institute and the H.E.G. lead to numerous publications both in the vascular and cardiac levels. The vascular medicine department has an Aixplorer® prototype with vascular and cardiac applications on site. The advantage of this technology is its ultrafastecho mode with very high temporal resolution which allows the vascular level to visualize and to calculate the speed of the arterial pulse wave which is correlated to the local rigidity.

The use of this innovative technique in aortic bicuspid will hopefully validate the evaluation of the carotid velocity of the pulse wave as an easily accessible prognostic marker of aortic dilation.

Purpose of the research

The objective is the development and validation of morphological markers informative of aortic dilatation in order to improve the precision of the risk of aneurysm of the thoracic aorta and of acute aortic syndrome for patients with BAV.

The primary objective of this study is to demonstrate a correlation between the aortic local PWV measured with MRI and the progression of the thoracic aorta diameters measured by MRI after a follow-up of 2 years

The secondary objectives are:

1. To demonstrate a correlation between the progression of the dilatation of the different segments of the thoracic aorta with the following measures:

   * Aortic distensibility measured in MRI at the Valsalva sinus and at the ascending tubular aortic level.
   * Aortic distensibility measured in TTE of the same segments in TM and in B mode .
   * Carotid pulse rate measured on carotid arteries by UF.
2. To demonstrate a correlation between the progression of the dilatation of the different segments of the thoracic aorta with the following environmental risk factors:

   * Active Smoking
   * Diabetes
   * Hypertension
   * Familial form of aortic BAV (defined by the presence of a relative, 1st or 2nd degree, with BAV or thoracic aortic aneurysm)
   * Morphological type of BAV
   * Aortic coarctation

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age,
* confirmed BAV by TTE computed tomography or MRI.
* Adults benefiting from a social security scheme,
* having received information on the research
* having signed the consent form

Exclusion Criteria:

* Patient with a syndromic form of BAV:
* Loeys-Dietz syndrome,
* Turner syndrome
* Williams-Beuren syndrome
* Shone syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Evaluation of the progression of artic dilation with MRI | For each patient, inclusion in the study will be associated with one-day hospitalization with: MRI (=first MRI), TTE and UF (at T0). Patients will then be re-examined after 2 years to perform a second MRI to assess aortic dilatation (T=2 years).
  The measure evaluates a change, which is why there is more than one time point. For patients, a first MRI and a second MRI will be performed after 2 years (+/- 2 months) in order to evaluate prospectively the progression of aortic dilatation according to stiffness parameters.

SECONDARY OUTCOMES:
Comparison of aortic stiffness evaluation with different methods TTE, MRI, UF | For each patient, inclusion in the study will be associated with one-day hospitalization with: MRI (=first MRI), TTE and UF (at T0). Patients will then be re-examined after 2 years to perform a second MRI to assess aortic dilatation (T=2 years).
  Comparison of aortic stiffness evaluation with different methods TTE, MRI, UF

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel MESSAS, Principal Investigator — APHP
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: No